CLINICAL TRIAL: NCT03736317
Title: Evaluation of the Effect of Repetitive Transcranial Magnetic Stimulation in Craving in Methamphetamine Use Disorder
Brief Title: Transcranial Magnetic Stimulation for Treatment of Methamphetamine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MZhao-009
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Amphetamine Use Disorders
Keywords: Amphetamine-type stimulants; prefrontal-striatal circuits; rTMS; individualized therapy; craving; relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Sham Comparator): Sham TBS delivered on left dlPFC or medial prefrontal cortex of amphetamine-dependent patients. Stimulation pulses are the same as the real group.
  Interventions: Device: sham TBS
- real mPFC cTBS group (Experimental): The real cTBS stimulation pattern will be delivered on the medial prefrontal cortex.
  Interventions: Device: real mPFC cTBS
- real dlPFC iTBS group (Experimental): The real iTBS stimulation pattern will be delivered on the left dorsal prefrontal cortex.
  Interventions: Device: real dlPFC iTBS
- real dlPFC iTBS + real mPFC cTBS group (Experimental): Combination therapy of real iTBS stimulation delivered on the left dorsal prefrontal cortex and real cTBS stimulation delivered on the medial prefrontal cortex.
  Interventions: Device: real dlPFC iTBS + real mPFC cTBS

INTERVENTIONS:
Device: sham TBS — Stimulate the dorsal lateral prefrontal cortex or medial prefrontal cortex for 2 weeks by sham Theta-burst stimulation (TBS), five times for a week with the sham coil.
  Arms: control group
Device: real mPFC cTBS — Stimulate the medial prefrontal cortex with the cTBS pattern. The therapy will be conducted for 2 weeks and five times for a week.
  Arms: real mPFC cTBS group
Device: real dlPFC iTBS — Stimulate the dorsal lateral prefrontal cortex with the iTBS pattern. The therapy will be conducted for 2 weeks and five times for a week.
  Arms: real dlPFC iTBS group
Device: real dlPFC iTBS + real mPFC cTBS — Stimulate the dorsal lateral prefrontal cortex with the iTBS pattern, and stimulate medial prefrontal cortex with the cTBS pattern. The therapy will be conducted for 2 weeks and five times for a week.
  Arms: real dlPFC iTBS + real mPFC cTBS group

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) was used to treat methamphetamine use disorder in previous studies, while the evidence-based protocols still required. The aim of this research is to develop more applicable rTMS intervention pattern and protocols to reduce craving and relapse of methamphetamine-dependent patients.

DETAILED DESCRIPTION:
The limbic circuit and executive control circuit are two important frontal-striatal neural circuits associated with drug dependence. Previous studies showed increased functional activity within the limbic neural circuit (e.g. medial prefrontal cortex (mPFC) and ventral striatum) in the presence of a salient cue and decreased activity in the executive control circuit (e.g. dorsal prefrontal cortex and dorsal striatum). TMS was used to reverse the activities of these two circuits, by using continuous TBS and intermittent TBS, respectively. In this study, vmPFC cTBS was conducted to modulating the limbic circuit, while left dlPFC iTBS was conducted to modulating the executive control circuit. Combined treatment of vmPFC cTBS and left dlPFC iTBS was conducted to modulating two circuits simultaneously. Focused on evaluating the efficacy of the interventions and investigate the mechanisms, neuropsychological tests, biochemical tests, and electroencephalography will be used to investigate the neurobiological mechanism of the methamphetamine use disorder, craving, and relapse. The study will be very helpful to develop evidence-based rTMS protocols for methamphetamine-dependent patients in clinical practice and decrease harm for both the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
* Primary school degree or above
* Normal vision and hearing
* Dextromanual
* Less than one month before last drug use

Exclusion Criteria:

* Have a disease that affect cognitive function such as history of head injury, cerebrovascular disease, epilepsy, etc
* Have cognitive-promoting drugs in the last 6 months
* Other substance abuse or dependence in recent five years (except nicotine)
* Mental impairment, Intelligence Quotient (IQ) < 70
* Mental disorders
* Physical disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale | 12 months.
  evaluate all participants' craving for for methamphetamine assessed by Visual Analog Scales (VAS). Score of VAS range from 0 to 10, and higher values represent high level of craving.

SECONDARY OUTCOMES:
Number of participants who relapse | 12 months
  Follow up with patients after discharge, evaluate number of participants who relapse
Depression status assessed by Patient Health Questionnaire-9(PHQ-9) | 12 months
  evaluate all participants' depression status by Patient Health Questionnaire-9(PHQ-9), PHQ-9 range from 0 to 27, and higher values represent more severe level of depression.
Anxiety status assessed by Generalized Anxiety Disorder Screener (GAD-7) | 12 months
  evaluate all participants' anxiety status by Generalized Anxiety Disorder Screener (GAD-7). PHQ-9 range from 0 to 21, and higher values represent more severe level of anxiety.
Cognitive function assessed by CogState Battery (CSB) | 12 months
  evaluate all participants' cognitive function by the computerized CogState Battery (CSB) Chinese version
Response inhibition function | 12 months
  assessed by Go nogo task under the electroencephalogram recording
Cue reactivity | 12 months
  assessed by Cue reactivity task under the electroencephalogram recording

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Compulsory Rehabilitation Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen T, Su H, Li R, Jiang H, Li X, Wu Q, Tan H, Zhang J, Zhong N, Du J, Gu H, Zhao M. The exploration of optimized protocol for repetitive transcranial magnetic stimulation in the treatment of methamphetamine use disorder: A randomized sham-controlled study. EBioMedicine. 2020 Oct;60:103027. doi: 10.1016/j.ebiom.2020.103027. Epub 2020 Sep 25. PMID 32980696